CLINICAL TRIAL: NCT05895591
Title: Exploratory Study to Assess Clinical and Biological Anti-aging Efficacy of a Cosmetic Cream in Women After 2 Months of Daily Use, Under Dermatological Control
Brief Title: Clinical and Biological Anti-aging Efficacy of a Cosmetic Cream
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RV4981A20210184
Record Dates: First submitted 2023-05-19; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-04

CONDITIONS: Anti-aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated Group (Experimental): all subjects will apply the study product
  Interventions: Other: Anti-aging cosmetic care product

INTERVENTIONS:
Other: Anti-aging cosmetic care product — * frequency of application: Once a day (in the morning)
  * modalities of application: Apply the cream on face (according to normal conditions of use) and on treated forearm, massage until complete penetration
  * area: The whole face, neck, neckline and one randomized forearm (external photo-exposed area) the other forearm is untreated
  * duration of investigational product application: 56 days (a window of + 72 hours is allowed)
  * quantity: 2 pressures of product for the whole face, neck and neckline and 1 pressure of product for the treated forearm

SUMMARY:
The aim of the study is to determine the efficacy of the investigational product "Cream " :

* on skin network after 56 days of daily application
* on biological parameters linked to cellular communication involved in senescence
* on sebum composition (metagenomics and metabolomics analysis)

DETAILED DESCRIPTION:
This study will be conducted as a monocentric, randomized (for side of product application on forearms), open trial.

4 visits are planned:

* Visit 1 - Inclusion (D1)
* Visit 2 - Follow-up visit (D29), a window of +72 hours is allowed for this evaluation,
* Visit 3 - End of the application period (D57), a window of +72 hours is allowed for this evaluation
* Visit 4 - Follow-up visit (D7 post-biopsies +/- 24h)

For a subject completing the study, the theoretical investigational product application will be 56 consecutive days up to 59 days maximum.

The study duration for each subject will be 67 days maximum.

ELIGIBILITY:
Inclusion Criteria:

* sensitive skin (declaratory judgment)
* face skin type: combination to normal skin
* presenting wrinkles and/or finelines on the whole face
* displaying saggy skin on the face (loss of firmness)
* presenting a lack of skin radiance, dull complexion and an inhomogeneous skin on the face

Exclusion Criteria:

Related to the treatment/product:

* having had any surgery, chemical or significant invasive dermo-treatment on the experimental area considered by the Investigator liable to interfere with the study data
* having undergone techniques with aesthetic aim on study areas (chemical peel, mechanical dermabrasion, laser, pulsed flash lamp etc.) or having made injections of anti-wrinkle products (collagen, hyaluronic acid, botulinic toxin etc.)
* having applied products with an anti-aging action (Retinoic acid, retinol, retinaldehyde, A.H.A. etc.)

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Assessment of skin network (SRa parameter) by Fringe projection on silicone rubber replica (on one randomized forearm) | Change from baseline to Day 57
  SRa: Average roughness (mm). Average variations in amplitude of the relief integrated into the studied surface.
Assessment of skin network (SRq parameter) by Fringe projection on silicone rubber replica (on one randomized forearm) | Change from baseline to Day 57
  SRq: Roughness with regards to the average quadratic plan (mm).
Assessment of sebum metabolites' composition | Change from baseline to Day 57
  Metabolomics analysis from sebum samples using mass spectrometry
Assessment of skin metagenomic composition | Change from baseline to Day 57
  Metagenomics analysis from sebum samples using targeted DNA sequencing
Expression of cellular communication markers linked to senescence | Day 57
  RNA expression from skin biopsies using RNA-Seq

CONTACTS AND LOCATIONS:
Locations (1):
- Spincontrol, Tours, France